CLINICAL TRIAL: NCT01487486
Title: Proteomics & Glyco-Proteomic Analysis of Follicular Fluid Derived From Health Patient/Donors and Polycystic Ovary Syndrome Patients
Brief Title: Proteomics & Glyco-Proteomic Analysis of Follicular Fluid
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Steven Lindheim, Professor, University of Cincinnati
Other Study IDs: Proteomics of FF in PCOS
Record Dates: First submitted 2011-11-16; First posted 2011-12-07 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Polycystic Ovary Syndrome; Normal Volunteers
Keywords: Polycystic Ovary Syndrome; PCOS; Follicular Fluid; Proteomics; Glyco-proteomics
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Follicular Fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal patients: Women with infertility diagnosis of male factor only or women who are oocyte donors
  Interventions: Drug: IVF Antagonist Protocol
- Polycystic Ovary Syndrome, High BMI: Women with Polycystic Ovary Syndrome with a BMI between 30-35
  Interventions: Drug: IVF Antagonist Protocol
- Polycystic Ovary Syndrome, Low BMI: Women with Polycustic Ovary Syndrom with a BMI between 20 & 25
  Interventions: Drug: IVF Antagonist Protocol

INTERVENTIONS:
Drug: IVF Antagonist Protocol — 1. Ovulation Induction: Achieved with recombinant FSH (Follistim®) with or without HMG (Menopur®) at total doses of 75-450 IU/day subcutaneous (SC) for 9-14 days.
  2. Ovulation Suppression: GnRH Antagonist (Ganirelix® - 250microgram 0.5ml) will be initiated following ovulation induction when lead follicle >14mm diameter on ultrasound and continued through the day of hCG (Novirel® or Ovidrel ®) injection
  3. hCG Injection: Once patient has met criteria for oocyte retrieval, she will inject either Novarel® (5,000-10,000 units Intramuscular) or Ovidrel® (250microgram - 500microgram SC) 35 hours prior to oocyte retrieval.

SUMMARY:
To the best of the investigators knowledge, exhaustive characterization of the low and high abundant proteins and glyco-proteins of the Follicular Fluid (FF) has not yet been achieved. Such an analysis may provide critical molecular data on the role of the FF in oocyte maturation and may identify specific changes in the FF proteome of patients with gynecologic problems, such as Polycystic Ovary Syndrome (PCOS).

Specific Aims

1. To perform a comprehensive analysis of normal human FF using sensitive mass spectrometry in combination with conventional approaches for proteomic evaluation and using HPLC and Western blot for glyco-proteomic analysis.
2. Characterize differential proteomic and glyco-proteomic patterns of the FF in normal women compared to lean and obese women with PCOS.
3. To supplement the differential proteomic and glyco-proteomic analysis with steroid hormone analysis in all FF samples.

DETAILED DESCRIPTION:
In this study, we plan to utilize ultrasensitive mass spectrometry (MS) and other conventional proteomic approaches to identify the low and high abundant proteins present in human FF. Additionally, we plan to use high-performance liquid chromatography (HPLC) and Western blot techniques to evaluate the Neu5Gc and glycan array based ELISA techniques to detect anti-Neu5Gc antibody profile in human FF. This analysis will be performed on FF samples obtained from normal women undergoing In-Vitro Fertilization and Embryo Transfers (IVF-ET) for a male factor alone and oocyte donors from our 3rd Party Reproduction Program and from lean and obese women with PCOS. This study will provide information on protein, glycoprotein, and steroid hormone expression during normal folliculogenesis and during the pathologic condition of PCOS, which should also provide basic scientific information on normal and abnormal oocyte development.

Human FF bathes the developing oocyte. Previous studies indicate that the FF contains cytokines, steroidal and protein hormones, and growth factors. The presence of proteins with such significant biological properties implies a paracrine and autocrine role for the FF in promoting normal oocyte development. Furthermore, the presence of any antigenic sialic acid Neu5Gc and the presence of antibodies targeting these antigenic glycoconjugates (glycolipid and glycoproteins decorated with sialic acid) may interfere with oocyte development, hormonal expression, fertilization, and possibly implantation. Here we hypothesize that an exhaustive proteomic and glyco-proteomic characterization of human FF is essential for a thorough understanding of its biological significance. We also hypothesize that PCOS may have differential expression of the FF protein and glyco-protein milieu, and that the expression may differ further between lean and obese women with PCOS. PCOS represents a heterogeneous disorder. The severity of hyperandrogensim, metabolic and menstrual disturbance, and obesity is variable with up to 40% not clinically expressing signs of classic hyperandrogenism. On the other hand, these atypical, often lean, PCOS women can have impaired glucose tolerance and diabetes. Reports suggest that these lean PCOS women have altered serum IGFBP-1, a characteristic endocrine feature of patients with obese PCOS, and related to hyperinsulinemia and/or obesity. The lean phenotype of PCOS and its significance is unclear but may represent a cryptic or unexpressed form of PCOS or may be a prelude to individuals who will later manifest clinical signs of obese/overweight PCOS. Changes in expression may be expected because of the different amounts of steroidal hormones and inflammatory markers in the FF derived from women with PCOS.

ELIGIBILITY:
Inclusion criteria: Inclusion Criteria All

1. Female patients undergoing controlled ovarian hyperstimulation (COH), transvaginal oocyte aspiration (TVA), and Saline Infused Sonography (SIS) with UL collection
2. Age <35 y/o at time of in vitro fertilization (IVF) cycle
3. Normal ovarian function defined Day 3 Follicular Stimulating Hormone (FSH) <8 pg/ml or Anti-Mullerian Hormone (≥ 1.0 ng/ml)

Inclusion Criteria Controls:

1. Female patients undergoing COH and TVA donating her oocytes
2. Female patients undergoing COH and TVA for male factor infertility only (i.e. no female causes of infertility)
3. Normal menstrual cycles

Inclusion Criteria Lean PCOS:

1. Diagnosis of PCOS by Rotterdam Criteria
2. BMI ≤ 25 kg/m2 Inclusion Criteria Classic PCOS

1. Diagnosis of PCOS by Rotterdam Criteria 2. BMI > 30 kg/m2

Exclusion criteria:

1. Age ≥ 35 y/o
2. Female partners with infertility associated diagnosis (i.e. tubal factor, cervical factor, endometriosis)
3. Unexplained infertility

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing In Vitro Fertilization who have:
  1. male factor only infertility diagnosis or are oocyte donors
  2. PCOS
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Proteomic analysis | Participants will be followed for one IVF cycle including pregnancy outcomes, on average this will be 6-8 weeks.
  For proteomic analysis the follicular fluid samples will be either directly analyzed by MS or will be processed to deplete albumin which is likely to be present in very high abundance in the FF.

SECONDARY OUTCOMES:
Hormone analysis | Participants will be followed for one IVF cycle including pregnancy outcomes, on average this will be 6-8 weeks.
  An aliquot of FF from each patient will be analyzed for the following steroid hormones: progesterone, 17-alpha-hydroxyprogesterone, androstenedione, testosterone, estradiol, and dihydrotestosterone.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lindheim, MD, MMM, Principal Investigator — University of Cincinnati
Locations (1):
- Center for Reproductive Health, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Farquhar CM, Birdsall M, Manning P, Mitchell JM, France JT. The prevalence of polycystic ovaries on ultrasound scanning in a population of randomly selected women. Aust N Z J Obstet Gynaecol. 1994 Feb;34(1):67-72. doi: 10.1111/j.1479-828x.1994.tb01041.x. PMID 8053879
- [Background] Carmina E, Lobo RA. Do hyperandrogenic women with normal menses have polycystic ovary syndrome? Fertil Steril. 1999 Feb;71(2):319-22. doi: 10.1016/s0015-0282(98)00455-5. PMID 9988405
- [Background] Carmina E, Wong L, Chang L, Paulson RJ, Sauer MV, Stanczyk FZ, Lobo RA. Endocrine abnormalities in ovulatory women with polycystic ovaries on ultrasound. Hum Reprod. 1997 May;12(5):905-9. doi: 10.1093/humrep/12.5.905. PMID 9194637
- [Background] Clayton RN, Ogden V, Hodgkinson J, Worswick L, Rodin DA, Dyer S, Meade TW. How common are polycystic ovaries in normal women and what is their significance for the fertility of the population? Clin Endocrinol (Oxf). 1992 Aug;37(2):127-34. doi: 10.1111/j.1365-2265.1992.tb02296.x. PMID 1395063
- [Background] Mendoza C, Ruiz-Requena E, Ortega E, Cremades N, Martinez F, Bernabeu R, Greco E, Tesarik J. Follicular fluid markers of oocyte developmental potential. Hum Reprod. 2002 Apr;17(4):1017-22. doi: 10.1093/humrep/17.4.1017. PMID 11925399
- [Background] Polson DW, Adams J, Wadsworth J, Franks S. Polycystic ovaries--a common finding in normal women. Lancet. 1988 Apr 16;1(8590):870-2. doi: 10.1016/s0140-6736(88)91612-1. PMID 2895373
- [Background] Suikkari AM, Koivisto VA, Rutanen EM, Yki-Jarvinen H, Karonen SL, Seppala M. Insulin regulates the serum levels of low molecular weight insulin-like growth factor-binding protein. J Clin Endocrinol Metab. 1988 Feb;66(2):266-72. doi: 10.1210/jcem-66-2-266. PMID 2448329
- [Background] Conover CA, Lee PD, Kanaley JA, Clarkson JT, Jensen MD. Insulin regulation of insulin-like growth factor binding protein-1 in obese and nonobese humans. J Clin Endocrinol Metab. 1992 Jun;74(6):1355-60. doi: 10.1210/jcem.74.6.1375600.